CLINICAL TRIAL: NCT02470832
Title: A Study to Investigate the Effect of CYP3A Inhibition on the Pharmacokinetics of RG1662 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: WP29402; 2015-000261-31 (EudraCT Number)
Record Dates: First submitted 2015-05-13; First posted 2015-06-12 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Healthy Patient Study
MeSH Terms: interventions — Itraconazole

ARMS (3):
- Combination therapy RG1662 + itraconazole (Experimental): Days 20-29: Oral administration RG1662 twice daily within 30 minutes of a meal + 2 x 100 mg itraconazole once daily with food
  Interventions: Drug: RG1662; Drug: itraconazole
- RG1662 Monotherapy (Experimental): Days 1-10: RG1662 120 mg twice daily (b.i.d.) within 30 minutes of a meal for 10 days (Days 1 to 9, Day 10 only a.m. dose). (Cohort A subjects will receive 1 x 120 mg RG1662 tablets twice daily. In Cohorts B and C the dose of RG1662 will be decided upon following review of the interim safety and pharmacokinetic data of the 4 subjects in Cohort A.)
  Interventions: Drug: RG1662
- itraconazole Monotherapy (Experimental): Days 15-19: 200 mg of itraconazole twice daily for 5 days (Days 15 to 18, Day 19 only a.m. dose)
  Interventions: Drug: itraconazole

INTERVENTIONS:
Drug: RG1662
  Arms: Combination therapy RG1662 + itraconazole; RG1662 Monotherapy
Drug: itraconazole
  Arms: Combination therapy RG1662 + itraconazole; itraconazole Monotherapy

SUMMARY:
The study is being conducted to investigate the effect of itraconazole treatment in the pharmacokinetics of RG1662. It is also to evaluate the exposure of RG1662 vs. QTc response relationship and the safety and tolerability of RG1662 when given in combination with itraconazole in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers
* Ages 18 to 60 years, inclusive
* A body mass index (BMI) between 18 to 32 kg/m2, inclusive
* Agreement to comply with study restrictions

Exclusion Criteria:

* History of epilepsy, convulsions or significant head injury or electroencephalogram (EEG) abnormalities
* Electrocardiogram (EGC) or vital signs abnormalities
* Significant history of drug allergy, as determined by the Investigator, or a known hypersensitivity to any of the ingredients of any of the study treatments
* Use of any drugs or substances that are known to be substrates, inducers or inhibitors of CYP3A4 within 30 days of the first dose administration
* Pregnant or lactating
* Any other clinically relevant abnormalities, concomitant diseases or ongoing medical conditions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from 0-t (AUC0-t) | Within 29 days
Maximum observed plasma concentration (Cmax) | Within 29 days
Time to maximum observed plasma concentration (Tmax) | Within 29 days

SECONDARY OUTCOMES:
Change from baseline in QTcF | Up to 29 days
Incidence of adverse events | Within 43 days
Clinically significant changes from baseline in physical examination or laboratory parameters | Within 29 days
Mean model parameters of RG1662 concentration vs. QTcF changes | Within 29 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Leeds, United Kingdom